CLINICAL TRIAL: NCT04364906
Title: Comparison of the Effects of Quadratus Lumborum Block 2 and 3 (QLB 2 and QLB 3) on Post-operative Analgesia in Cesarean Section Surgery
Brief Title: Comparison of the Effects of QLB 2 and QLB 3 on Post-operative Analgesia in Cesarean Section Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Caner Genç, Medical Doctor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: QL20011990
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Analgesia; Acute Pain; Chronic Pain
Keywords: Regional Anesthesia; Acute and chronical pain; Quadratus Lumborum Blocks; Cesarean Section; Spinal Anesthesia
MeSH Terms: conditions — Agnosia; Acute Pain; Chronic Pain | interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: Randomization of the study will be done by a doctor who will not participate in patient follow-up with closed envelopes using computer generated randomization codes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesia doctor who will perform the interfascial plane block (QLB 2, 3) will be informed with a sealed envelope by an independent assistant outside the study, and the patient will not know which block is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block 2 (Active Comparator): Quadratus Lumborum Block 2 (QLB 2) will be performed the patients in Group A after the cesarean section surgery. Patient controlled analgesia device (PCA) is used for all the patients in the first 24 hours postoperatively
  Interventions: Other: Regional anesthesia
- Quadratus Lumborum Block 3 (Active Comparator): Quadratus Lumborum Block 3 (QLB 3) will be performed the patients in Group B after the cesarean section surgery. Patient controlled analgesia device (PCA) is used for all the patients in the first 24 hours postoperatively
  Interventions: Other: Regional anesthesia

INTERVENTIONS:
Other: Regional anesthesia — The effects of QLB 2, 3 interfascial plane blocks on post-operative analgesia after cesarean section surgery
  Other Names: Quadratus Lumborum Block 2; Quadratus Lumborum Block 3

SUMMARY:
This study evaluates the post-operative analgesic effects of quadratus lomborum block 2 and 3 (QLB 2, 3) in patients having cesarean section with spinal anesthesia. Spinal anesthesia will be performed to all patients for the surgery.

DETAILED DESCRIPTION:
In this study, patients are divided into two groups. After the spinal anesthesia is performed and cesarean section surgery is over; QLB 2 block will be performed to patients in Group A ; while QLB 3 block will be performed to patients in Group B.

In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively.

Group A - Patients in group A will have QLB 2 block after the surgery. In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively.

Group B - Patients in group B will have QLB 3 block after the surgery. In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant for at least 37 weeks
* Planning an elective cesarean operation
* Being between the ages of 18-45

Exclusion Criteria:

* ASA 3-4 patients with comorbitidies (Serious renal, cardiac, hepatic disease)
* Being operated with general anesthesia
* Obesity (> 100 kg, BMI> 35 kg / m2)
* Contraindication of regional anesthesia (quagulopathy, abnormal INR, thrombocytopenia, infection at the injection site)
* Hypersensitivity to local anesthetics or a history of allergy
* Patients with a history of opioid use longer than four weeks
* Patients with psychiatric disorders
* Patients with anatomic deformity
* Patients who do not want to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women planned for elective cesarean operation
Enrollment: 80 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the first 24 hours after surgery | 1 day
  Morphine consumption in the first 24 hours will be counted by IV patient controlled analgesia device (PCA). Patients will be able to request opioids via PCA device when the nrs score is above 4.

SECONDARY OUTCOMES:
Post-operative acute pain | 1 day
  Pain status will be evaluated based on NRS scores. Pain status will be evaluated at 1, 3, 6, 9, 12, 18, 24. hours after surgery. Each NRS is scores 0-10. (0=no pain ; 10=pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: ERSİN KÖKSAL, MD, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Other, Turkey (Türkiye)